CLINICAL TRIAL: NCT01641627
Title: Phase 2 Randomized Clinical Trial, Efficy of a Proprioceptive Stimulation Device in Term of Prevention of Muscle Atrophy of the Calf After Total Knee Replacement
Brief Title: Preventive Effect of Proprioceptive Stimulation on Muscle Atrophy
Acronym: PrevAtrophy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010_05; 2011-A0031-40 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2012-05-22; First posted 2012-07-17 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Knee Arthritis
Keywords: knee arthritis; muscle atrophy; proprioceptive stimulation; vibrations
MeSH Terms: conditions — Muscular Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- vibration (Experimental): proprioceptive stimulation of the lower limb using vibration and plantar pressure boots
  Interventions: Procedure: proprioceptive stimulation

INTERVENTIONS:
Procedure: proprioceptive stimulation — tendon vibrations and plantar stimulation with a therapeuthic orthosis, 4x30 min/day during 14 days
  Other Names: therapeutic boots, vibration boots

SUMMARY:
Confinement to bed, which occurs in many pathological situations, induces a muscle atrophy and a loss of muscle strength. Muscle atrophy is associated to impaired performance in motor tasks, such as posture and locomotion, and is therefore a major cause of loss of autonomy. It requires a stay in follow-up and rehabilitation service, and thus lengthens the duration of hospitalisation.

Data underline the importance of afferent input integrity in the maintenance of muscle characteristics and postural control, and suggest that countermeasure programs based on the stimulation of proprioceptive inputs could be efficient to prevent muscle atrophy and falls. In particular, fundamental studies performed in rodents by the investigators laboratory have demonstrated that the adverse structural and functional adaptations which occur during muscle deconditioning can be counteracted through adequate physiological stimuli such as activation of proprioceptors. Based on this scientific expertise, the investigators aim is thus to prevent muscle atrophy and its functional consequences on posture and locomotion, following a surgical intervention in humans .

The investigators will develop a device allowing stimulation of foot and ankle proprioceptors. In order to facilitate the evaluation of its efficiency, the device will be tested on a selected population confined to bed during a post-operative period (knee replacement). It efficiency will be evaluated by means of three parameters: muscle force of ankle plantar flexor, muscle volume of lower limb muscles, functional outcome (gait and balance analysis).

The technique developed in the present project could bring benefits to patients confined to bed, or in elderly. Preventing or retarding development of muscle atrophy will beneficiate to health and quality of life of these patients. In addition, this device might allow to consider therapeutic strategies for prevention of atrophy in neuromuscular pathologies.

DETAILED DESCRIPTION:
The aim of the study is to study the efficacy of a proprioceptive stimulation device on prevention of calf muscle atrophy after a total knee replacement.

The investigators developped a safe vibration and pressure stimulation device for le lower limb. The investigators want to carry out a RCT in order to demonstrate the efficacy of the stimulation device, compared to a not stimulated controle group.

ELIGIBILITY:
Inclusion Criteria:

* patients waiting for knee replacement

Exclusion Criteria:

* neurologic disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-03; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
The Isokinetic Maximal Voluntary strenght of the plantar floxors of the ankle. The outcome measure is assessed using an isokinetic strength assesment device (CON-TREX , CVM-AG, Switzerland) | 1.5 year
  The patients will perform series of maximal contraction of the plantar flexors against the lever arm of the isokinetic device at 3 different angular speeds : 180°/s 90°/s, 120°/sec

SECONDARY OUTCOMES:
Volume of the Soleus muscle | 1.5 years
  Ultrasound measurement of the soleus muscle volume

CONTACTS AND LOCATIONS:
Overall Officials: vincent TIFFREAU, MD-PhD, Principal Investigator — Univerity Hospital Lille 2
Locations (1):
- CHRU de Lille, Lille, Nord, France